CLINICAL TRIAL: NCT02381236
Title: G-202-005: An Open-Label, Single-Arm, Phase II Study to Evaluate the Safety and Activity of G-202 Administered in the Neoadjuvant Setting Followed by Radical Prostatectomy in Patients With Adenocarcinoma of the Prostate
Brief Title: G-202 in the Neoadjuvant Setting Followed by Radical Prostatectomy in Patients With Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GenSpera, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G-202-005
Record Dates: First submitted 2015-02-23; First posted 2015-03-06 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- G-202 (Experimental): G-202 administered by intravenous infusion on 3 consecutive days of a 28-day cycle
  Interventions: Drug: G-202

INTERVENTIONS:
Drug: G-202 — G-202 administered by intravenous infusion on Days 1, 2 and 3 of each 28-day cycle for up to 3 cycles
  Other Names: Mipsagargin

SUMMARY:
A single-arm, open-label Phase II clinical trial to evaluate the effect of G-202 on the perfusion and volume of the prostate using non-invasive multiparametric prostate magnetic resonance imaging (mpMRI).

DETAILED DESCRIPTION:
More than one-third of patients with localized high-risk prostate cancer who undergo radical prostatectomy eventually relapse with distant disease and some data suggest that neoadjuvant treatment in this patient population may be helpful. This study is based on prodrug tumor targeting, in which an inactive form of a toxic agent is administered systemically and gets activated in specific locations in the body, resulting in higher concentrations of the cytotoxic form at the tumor location. G-202 is a prodrug that is activated in prostate cancer tissue and in the blood vessels of tumors, but not normal tissue; once activated, G-202 leads to disruption of intracellular calcium levels and subsequent induction of apoptosis. Thus, G-202 is expected to bring about cell death in prostate cancer cells and to destroy the blood supply of prostate tumors. G-202 has led to disease stabilization in some patients, but the drug has not been evaluated in the neoadjuvant setting. This single-arm, open-label Phase II clinical trial will evaluate the safety and activity of G-202 in patients with localized high-risk prostate cancer prior to radical prostatectomy. Through its effects on the neovasculature of tumors, G-202 is anticipated to disrupt the blood supply of the prostate tumor, resulting in decreased perfusion and subsequent tumor volume. The primary endpoint of this study is evaluation of G-202 on the perfusion and volume of the prostate using non-invasive multiparametric prostate magnetic resonance imaging (mpMRI).

ELIGIBILITY:
Inclusion Criteria:

* ECOG Performance Status < 2
* Histological confirmation of prostatic adenocarcinoma that is confined to the prostate without evidence of regional and/or distant metastasis
* Clinical stage T1c or T2a with high-grade disease (Gleason 8-10) on initial biopsy, clinical stage T2b-T2c with Gleason grade 7 (4+3), or clinical stage T3
* Negative bone scan and CT of chest and abdomen within 6 weeks of first infusion of G-202
* Candidate for radical prostatectomy
* Adequate hematologic function (ANC ≥ 1200/mm3, hemoglobin ≥ 8.5 g/dL, platelets ≥ 75,000/mm3)
* Adequate hepatic function (albumin ≥ 2.8 g/dL, AST and ALT ≤ 5 x ULN, total bilirubin < 2 mg/dL)
* Adequate renal function (proteinuria level ≤ 2+, serum creatinine ≤ 1.5 x ULN)
* Acceptable coagulation profile (no history of substantial non-iatrogenic bleeding diatheses, INR ≤ 2.3, aPTT ≤ 1.5 x ULN)
* Ejection fraction (LVEF) ≥ 45% measured by echocardiogram
* Willing to use acceptable methods of contraception to avoid pregnancy

Exclusion Criteria:

* Prostatic adenocarcinoma with neuroendocrine differentiation or small cell features
* Unable to tolerate mpMRI
* Surgical resection or major surgery within 4 weeks or stereotactic biopsy within 1 week prior to first G-202 treatment
* Previous or current hormonal treatment, chemotherapy, radiation therapy, immunotherapy, or other investigational status drug for prostatic adenocarcinoma
* Currently requiring systemic administration of antibiotics or chronic administration of anti-viral agents
* Use of anti-coagulants is limited to local use for control of central line patency
* History or evidence of cardiac risk
* Uncontrolled cardiac or coronary artery disease
* Uncontrolled hypertension or hypertension requiring treatment with more than 2 anti-hypertensive agents
* Severe or uncontrolled medical disease
* Severe gastrointestinal bleeding within 12 weeks prior to treatment with G-202
* Known history of HIV, hepatitis B or hepatitis C
* Use of herbal products that may decrease PSA levels (e.g., saw palmetto) or systemic corticosteroids
* Documentation of keratosis follicularis
* Requirement for chronic use of medications known to be strong inhibitors or inducers of cytochrome (CYP3A4) iso-enzymes
* Another primary malignancy, except non-melanoma skin cancer, that has not been in remission for at least 2 years.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2016-02; Primary Completion 2016-12 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Volume of the prostate using multiparametric prostate magnetic resonance imaging (mpMRI) | 12 weeks from first administration of G-202
  mpMRI performed after 3 cycles of treatment prior to prostatectomy
Perfusion of the prostate using multiparametric prostate magnetic resonance imaging (mpMRI) | 12 weeks from first administration of G-202
  mpMRI performed after 3 cycles of treatment prior to prostatectomy

CONTACTS AND LOCATIONS:
Overall Officials: Robert Amato, D.O., Principal Investigator — University of Texas Health Sciences Center at Houston
Locations (1):
- University of Texas Health Sciences Center, Houston, Texas, United States